CLINICAL TRIAL: NCT05830136
Title: The Application of Sodium Bicarbonate Ringer's Solution on Perioperative Lactic Acid Concentration and Early Recovery Quality in Patients Undergoing Laparoscopic Hepatectomy
Brief Title: Application of Sodium Bicarbonate Ringer's Solution in Laparoscopic Hepatectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shijiang Liu, MD, Clinical Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-SR-386
Record Dates: First submitted 2023-02-27; First posted 2023-04-26 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Hepatic Ischemia
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Sodium bicarbonate Ringer's solution group
  Interventions: Drug: sodium bicarbonate Ringer's solution
- Group B (Active Comparator): Lactate Ringer's solution group
  Interventions: Drug: sodium bicarbonate Ringer's solution

INTERVENTIONS:
Drug: sodium bicarbonate Ringer's solution — Sodium bicarbonate Ringer's solution was used in Group A as intraoperative intravenous fluids. Lactate Ringer's solution was used in Group B as intraoperative intravenous fluids.
  Other Names: lactated Ringer's solution

SUMMARY:
Compared the effects of Sodium bicarbonate Ringer's solution and lactate Ringer's solution on the internal environment and hemodynamics of patients during laparoscopic liver resection, to observe the application prospect of sodium bicarbonate Ringer's solution in Laparoscopic hepatectomy.

DETAILED DESCRIPTION:
The study was a single-center prospective randomized controlled study. A total of 100 patients undergoing laparoscopic hepatectomy under general anesthesia were randomly divided into 2 groups: Group A, sodium bicarbonate Ringer's solution group(n=50); Group B, Lactate Ringer's solution group (intraoperative crystal fluid dilatation was lactate ringer's injection, n=50); Collect patients' arterial blood gas, blood pressure, heart rate, peripheral vascular resistance, heart rate, blood vessels, the active drug usage, 5% sodium bicarbonate injection usage, inflammation factors, transaminase, creatinine, etc. with the point of preoperative (T0), during liver specimens resected(T1), after liver specimens resected(T2), and the end of surgery (T3). Then statistical analysis and observe the application prospect of sodium bicarbonate Ringer's injection in Laparoscopic hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old,
2. patients who plan to undergoing laparoscopic hepatectomy ;
3. Willing to sign informed consent.

Exclusion Criteria:

1. age <18 years
2. pregnancy
3. active cardiac conditions (unstable coronary syndromes, decompensated heart failure, significant arrhythmias, severe valvular disease, history of congestive heart failure)
4. history of significant cerebrovascular disease
5. restrictive or obstructive pulmonary disease
6. uncontrolled hypertension
7. renal dysfunction (glomerular filtration rate <60 mL/min),
8. evidence of hepatic metabolic disorder (bilirubin >35 mmol/L)
9. presence of active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
lactic values | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 month.
  to compare the conditions of acid-base balance and internal environment between the two groups

SECONDARY OUTCOMES:
Amount of sodium bicarbonate injection (ml) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 month.
Value of pH | From the start of operation until the end of operation (during the operation).
Concentration of HCO3- | From the start of operation until the end of operation (during the operation).
Value of BE | From the start of operation until the end of operation (during the operation).
Concentration of Glucose | From the start of operation until the end of operation (during the operation).
Value of MAP | From the start of operation until the end of operation (during the operation).
Value of HR | From the start of operation until the end of operation (during the operation).
Concentration of CI | From the start of operation until the end of operation (during the operation).
Value of SVV | From the start of operation until the end of operation (during the operation).
Value of SVR | From the start of operation until the end of operation (during the operation).
Value of PPV | From the start of operation until the end of operation (during the operation).
Amount of norepinephrine | From the start of operation until the end of operation (during the operation).
Amount of phenylephrine | From the start of operation until the end of operation (during the operation).
Amount of ephedrine | From the start of operation until the end of operation (during the operation).
Amount of nitroglycerin | From the start of operation until the end of operation (during the operation).
Amount of milrinone | From the start of operation until the end of operation (during the operation).
Amount of furosemide | From the start of operation until the end of operation (during the operation).
time of palinesthesia from general anesthsia | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 month.
  postoperative palinesthesia, recovering time
time of stay in PACU | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 month.
extubation time | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 month.
Concentration of BUN | day 1 and day 3 after surgery.
Concentration of Cr | day 1 and day 3 after surgery.
Value of AST | day 1 and day 3 after surgery.
Value of ALT | day 1 and day 3 after surgery.
Amount of blood loss | intraoperative
  amount of blood loss during the operation.
Amount of blood transfusion | intraoperative
  amount of blood transfusion during the operation.
urinary output | intraoperative
  amount of urinary output during the operation.
15-item quality of recovery scale scores (QoR-15) | day 1 and day 3 after surgery.
  15-item quality of recovery scale scores. the minimum value is 0 and maximum value is 150, and whether higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Shijiang Liu, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Shijiang Liu, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No